CLINICAL TRIAL: NCT01676636
Title: Preference, Acceptability, and Palatability of Alternative Delivery Vehicles for Prenatal Calcium Supplementation Among Pregnant Women in Bangladesh
Brief Title: Delivery Vehicles for Prenatal Calcium Supplementation
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: The Sprinkles Global Health Initiative (Unknown); International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Principal Investigator, Stanley Zlotkin, Chief, Global Child Health, The Hospital for Sick Children
Other Study IDs: 1000032744
Record Dates: First submitted 2012-08-16; First posted 2012-08-31 (Estimated); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Pregnancy
Keywords: Pregnancy; Calcium; Supplements

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pregnant Women: Women who are 13 to 30 weeks pregnant. Each participant will take all 4 different calcium vehicles and decide which one they prefer.
  Interventions: Drug: Traditional Tablet; Drug: Chewable tablets; Drug: Unflavoured Powder; Drug: Flavoured Powder

INTERVENTIONS:
Drug: Traditional Tablet — The traditional tablets will be swallowed with liquid. Each tablet will contain 500 mg of calcium (as calcium carbonate), thus participants will be asked to take 3 per day.. Participants will be asked to take the tablets with a liquid of their choosing with a meal. Traditional tablets will function as a control in this study, as they represent what is widely available on the market in Bangladesh.
Drug: Chewable tablets — Chewable tablets are chewed in the absence of additional water. Each chewable tablet will contain 300 mg of calcium (as calcium carbonate), thus participants will be asked to take 5 per day. Participants will be asked to consume the chewable tablets with a meal.
Drug: Unflavoured Powder — The unflavoured powder with suspension agent will be tasteless and consumed by either adding it to a semi-solid food or drink of one's choosing. Appropriate foods for mixing with the powder will be at the discretion of the participants. This vehicle was selected on the basis that it would be easy to swallow, given the nausea associated with pregnancy. A similar product is Sprinkles, a multiple micronutrient powder developed at SickKids by Dr. Zlotkin.
Drug: Flavoured Powder — The flavoured powder with suspension agent will be consumed by adding it to clean water with a meal. This vehicle was also selected on the basis that it would be easy to swallow, given the nausea associated with pregnancy. Similar products include oral rehydration salts or artificial juice flavour crystals.

SUMMARY:
The SickKids-led research team is currently developing a prenatal micronutrient powder that will contain calcium, iron, and folic acid with different absorption characteristics. Once the powder is developed, it can be incorporated into various oral delivery vehicles. The overall effectiveness of a micronutrient program is highly dependent on the acceptance and regular consumption of supplements (i.e., adherence) by the targeted users. This is a study of the preference, acceptability, and palatability of 4 alternative delivery vehicles for the innovative prenatal multiple micronutrient supplement: traditional tablets, oral disintegrating tablets, unflavoured powder with a suspension agent, and flavoured powder with a suspension agent. This study will be conducted in Dhaka, Bangladesh. This study hypothesizes that that the formulation of the delivery vehicle will impact preference, acceptability, and palatability.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women ages 18 to < 40 years
* Gestational age of 13-30 completed weeks, estimated based on the recalled first day of the last menstrual period (LMP)
* Current residence in Dhaka at a fixed address
* Plan to remain in Dhaka for the duration of the study

Exclusion Criteria:

* Reported complications of current pregnancy
* Complicated medical or obstetric history that may increase the risk of preterm birth or prenatal complications, based on self-report
* Moderate or severe anaemia (hemoglobin < 90 g/L, accessed with Hemocue)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women who are between 13 and 30 weeks pregnant. Participants will be recruited from Shimantik .
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2012-10; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Frequency of Consumption of the Calcium Vehicle | Change from Baseline in Consumption of the Calcium Vehicle at day 22
  Consumption of the delivery vehicles will be measured during the once-weekly interactions with the research assistants in two ways: (1) by self-report from study participants; and (2) by counting the number of missing doses from those provided in the weekly supply.

SECONDARY OUTCOMES:
Acceptability | Day 1, Day 9, Day 16, Day 22
  Measured by colour, preparation, administration.
Ease of Use | Day 1, Day 9, Day 16, Day 22
  Measured by size and ease of swallowing.
Patibility | Day 1, Day 9, Day 16, Day 22
  Measured by taste, texture, aftertaste, and odour.

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Zlotkin, MD, Principal Investigator — The Hospital for Sick Children; Daniel Roth, MD, Principal Investigator — The Hospital for Sick Children
Locations (2):
- International Center for Diarrheal Disease Research, Dhaka, Bangladesh
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Baxter JA, Roth DE, Al Mahmud A, Ahmed T, Islam M, Zlotkin SH. Tablets are preferred and more acceptable than powdered prenatal calcium supplements among pregnant women in Dhaka, Bangladesh. J Nutr. 2014 Jul;144(7):1106-12. doi: 10.3945/jn.113.188524. Epub 2014 Apr 23. PMID 24759933